CLINICAL TRIAL: NCT02695888
Title: A Pilot Study of a Mobile Technology Monitoring System to Assess a Web-based Intervention for Teen Risky Driving
Brief Title: Mobile Technology Monitoring System to Assess a Web-based Intervention for Teen Risky Driving
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Collaborators: Children's Hospital of Philadelphia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 15-012431; 823913 (Other: University of Pennsylvania)
Record Dates: First submitted 2016-02-25; First posted 2016-03-01 (Estimated); Last update posted 2018-10-18 (Actual); Status verified 2018-03

CONDITIONS: Adolescent; Accidents, Traffic; Attention; Motor Vehicles

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Risky driving prevention (Experimental): Web-based behavioral intervention to promote teen driver attention to the roadway, addressing mobile technology and passengers.
  Interventions: Behavioral: Risky Driving Prevention
- Control group (Experimental): Web-based behavioral intervention for healthy lifestyles.
  Interventions: Behavioral: Teen Healthy Living

INTERVENTIONS:
Behavioral: Risky Driving Prevention — The web-based intervention to prevent risky driving targets knowledge, attitudes, perceived control and norms about driver inattention, with strategies to keep attention on the roadway.
  Other Names: Web-based intervention to prevent risky driving
  Arms: Risky driving prevention
Behavioral: Teen Healthy Living — The control group will receive a web-based intervention for general health promotion and is designed to enhance participants' knowledge and ability to reduce their risk of adverse health conditions including, obesity and heart disease.
  Arms: Control group

SUMMARY:
This research study examines the feasibility of using an in-vehicle mobile technology monitoring system to measure teen secondary task engagement during on-road driving as the outcome measure for a web-based intervention to prevent risky driving in novice teen drivers.

DETAILED DESCRIPTION:
This research study examines the feasibility of using an in-vehicle mobile technology monitoring system to measure teen secondary task engagement during on-road driving as the outcome measure for a web-based intervention to prevent risky driving in novice teen drivers. Approximately 20 teens who have been licensed for less than 90 days will be enrolled and evaluated at baseline, ~1 week and ~4 weeks. Participants will complete an intervention after the ~1 week assessment. This study will provide information on the feasibility of the web-based intervention to prevent risky driving and estimation of effect size of the intervention on cell phone use while driving.

ELIGIBILITY:
Inclusion Criteria:

1. Males or females age 16-17 years at time of enrollment (i.e. can turn 18 while enrolled in research and still be eligible).
2. Has their own iPhone 4S or newer or Android 4.3 or newer smartphone with data plan
3. PA driver's license for 90 days or less at time of teen assent
4. Personal email address and computer and internet access
5. Ability to read and write English
6. Primarily drives one vehicle with the ability to accommodate the DriveID device
7. Parental consent and teen assent

Exclusion Criteria:

1. Participation in a Center for Injury Research and Prevention at CHOP teen driving study within the past 6 months
2. Unable to follow study procedures

Ages: 16 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 28 (Actual)
Dates: Start 2016-03; Primary Completion 2016-12-29 (Actual); Study Completion 2016-12-29 (Actual)

PRIMARY OUTCOMES:
Retention of participants | Baseline (Study Visit 1) through approximately 1- month (Study Visit 4)
  Proportion of participants enrolled who complete Study Visit 1, Study Visit 2, Study Visit 3 and Study Visit 4.

SECONDARY OUTCOMES:
In-vehicle cell phone use | Baseline (Study Visit 1) through approximately 1- month (Study Visit 4)
  Difference between the intervention and control group on frequency of cell phone use while driving as monitored by an in-vehicle device
Self-reported driving behaviors | Baseline (Study Visit 1) through approximately 1- month (Study Visit 4)
  Difference between the intervention and control group on on self-report measures of driving behaviors

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - University of Pennsylvania, Philadelphia, Pennsylvania

IPD SHARING:
Plan to Share IPD: No